CLINICAL TRIAL: NCT06094621
Title: Effect of Pre-operative Virtual Visits on Care of Patients With Head and Neck Cancer Undergoing Surgery
Brief Title: Effect of Pre-operative Virtual Visits on Patients With Head and Neck Cancer Undergoing Surgery
Status: Withdrawn | Type: Observational
Why Stopped: No Investigator Interest
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCC 2023.067; HUM00236077 (Other: University of Michigan)
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-operative Visit Arm: Eligible participants for the interview and surveys will be those who have undergone a virtual visit by the head and neck surgery nurse practitioners before their scheduled surgical procedure.
  Interventions: Other: Survey
- No Pre-operative Visit Arm: Patients who also underwent surgical resection for head and neck cancer with free flap reconstruction at the University of Michigan through the Department of Otolaryngology but did NOT receive a pre-operative virtual visit. This cohort is a retrospective chart review study

INTERVENTIONS:
Other: Survey — For the patients who underwent a pre-operative virtual visit, data will be collected through semi-structured interviews conducted by trained research personnel. The interviews will be conducted in a one-on-one format, either in-person or via telephone, according to the participant's preference.
  Groups: Pre-operative Visit Arm

SUMMARY:
Patients with head and neck cancer often undergo complex surgeries requiring significant care post-operatively. This presents considerable psychosocial challenges in addition to their need to physically recover from a large surgery.

The study team will interview patients who have undergone virtual visits before their surgical procedures. The study aims to explore patients' experiences, satisfaction, and perceptions of virtual visits for informing and preparing them for surgery and their postoperative care needs.

The study team will also analyze the effects of the virtual visits on financial costs and patient outcomes such as length of hospital stay, delayed discharges due to social issues, and whether the virtual visits identified any significant medical concerns, etc. The study team will compare these to a randomly selected cohort of patients who also underwent surgical resection and reconstruction for head and neck cancer that did not get pre-operative virtual visits.

ELIGIBILITY:
Inclusion Criteria (Pre-operative Visit Arm)

* Patients > 18 years
* Underwent surgery for head and neck cancer with free flap reconstruction at the University of Michigan
* Underwent a pre-operative virtual visit.

Inclusion Criteria (NO Pre-operative Visit Arm)

* Patients > 18 years
* Underwent surgery for head and neck cancer with free flap reconstruction at the University of Michigan

Exclusion Criteria (Pre-operative Visit Arm)

* Patients who died within 60 days of surgery for head and neck cancer with free flap reconstruction at the University of Michigan.

Exclusion Criteria (NO Pre-operative Visit Arm)

* Patients who died within 60 days of surgery for head and neck cancer with free flap reconstruction at the University of Michigan.
* Patient underwent a pre-operative virtual visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be adult patients aged 18 and over who underwent surgical resection for head and neck cancer with free flap reconstruction at the University of Michigan through the Department of Otolaryngology.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of virtual visits as determined by satisfaction scores | at time of enrollment
  To examine the satisfaction scores of patients who undergo pre-operative virtual visits. The satisfaction scale is graded on a modified Likert scale. The endpoint for this primary objective is the score given by the patient on the interview-based survey

SECONDARY OUTCOMES:
Comparison in hospitalization between cohorts | up to 60 days after the surgical resection
  To examine if patients who undergo pre-operative virtual visits have reduced hospital length of stay (i.e. number of days hospitalization post-operatively) compared to patients who did not undergo these visits.
Comparison in post-operative communication | up to 60 days after the surgical resection
  To examine if patients who undergo pre-operative virtual visits have reduced post-operative communication measured in portal messages and phone calls compared to patients who did not undergo these visits.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Casper, Principal Investigator — University of Michigan

IPD SHARING:
Plan to Share IPD: No